CLINICAL TRIAL: NCT05267041
Title: Prospective Longitudinal Cohort Associated to Blood Collection, Pathological Samples Collection, and Radiological and Pathological Imaging Collection
Brief Title: Joint Thoracic Oncology Research Unit of LYon: Lung cancerS DatabaSE (ULYSSE)
Acronym: ULYSSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 69HCL21_1175
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Data collection; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: One questionnaire between diagnostic annoucement and first line treatement One 6 months later One before second line treatment One 6 months later after second line treatment Optionnal Veinous Blood Sample (28 mL) between the diagnostic annoucement and the first line of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of Adults with lung cancer (Experimental): Patients newly diagnosed with lung cancer.
  Interventions: Biological: Blood sample; Other: Questionnaire

INTERVENTIONS:
Biological: Blood sample — One optional veinous blood sampling (24 ML) between the first diagnostic annoucement and before the first treatment for lung cancer
Other: Questionnaire — to collect data not reported in the patient's medical file, such as passive smoking, family history of cancer, and attempts to quit smoking.

SUMMARY:
Prospective longitudinal cohort associated to blood collection, pathological samples collection, and radiological and pathological imaging collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for a thoracic cancer in the Lyon University Hospital: non-small cell lung cancer, small cell lung cancer, mesothelioma…
* Diagnosis can be done:

  * By cytology or pathologic assessment
  * Or by multidisciplinary team meeting decision:

    * Irradiation without morpho-metabolic sampling
    * Treatment without sampling based on non-invasive molecular data

Exclusion Criteria:

- Refusal to participate

For optional blood sampling :

* < 30 kg for blood collection
* No blood sampling schedule for care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2032-05-05 (Estimated); Study Completion 2042-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants registered in the lung cancer database | 20 years
  cohort open to recruitment during 10 years with 10 years of patients follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France